CLINICAL TRIAL: NCT00020189
Title: A Phase II Trial of Daily Bolus Flavopiridol for Five Consecutive Days in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Flavopiridol in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068028; NCI-00-C-0128; MB-401; NCI-T99-0066; NCT00005670 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2004-08

CONDITIONS: Head and Neck Cancer; Thromboembolism
Keywords: thromboembolism; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thromboembolism; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Aspirin; alvocidib; Clopidogrel

INTERVENTIONS:
Drug: acetylsalicylic acid
Drug: alvocidib
Drug: clopidogrel bisulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of flavopiridol in treating patients who have recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the standard response rate (complete response and partial response) and duration of response in patients with recurrent or metastatic squamous cell carcinoma of the head and neck treated with flavopiridol.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the effects of anti-platelet agents, aspirin and clopidogrel bisulfate, on the pharmacology of flavopiridol in these patients.
* Determine the effects of prophylactic anticoagulation with anti-platelet agents, aspirin and clopidogrel bisulfate, on the incidence of flavopiridol-related thrombosis in these patients.

OUTLINE: Patients receive flavopiridol IV over 1 hour on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients also receive oral aspirin and clopidogrel bisulfate beginning on day 0 and continuing throughout the study.

Patients are followed until death.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 1-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven squamous cell carcinoma of the head and neck

  * Metastatic disease at diagnosis OR
  * Persistent, metastatic, or recurrent disease after prior definitive surgery and/or radiotherapy
* No undifferentiated and nonkeratinizing carcinomas, including lymphoepitheliomas of all locations
* No nasopharynx tumors
* Bidimensionally measurable disease

  * Patients whose only measurable disease is within a prior radiotherapy port must have clearly progressive disease
* No metastatic or leptomeningeal CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* Absolute granulocyte count greater than 1,500/mm^3

Hepatic:

* See Other (Prior/Concurrent Therapy)
* SGOT and SGPT less than 2.5 times normal
* Bilirubin less than 1.5 times normal
* No history of hypercoagulopathies (e.g., protein C deficiency, protein S deficiency, or lupus anticoagulant)

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* Calcium no greater than normal
* No hypercalcemia refractory to bisphosphonates

Cardiovascular:

* No unstable or newly diagnosed angina pectoris
* No myocardial infarction within the past 6 months
* No class II-IV congestive heart failure
* No history of symptomatic carotid disease
* No concurrent asymptomatic carotid artery occlusion (70% or greater) in one or both arteries by Doppler ultrasound
* No symptomatic atherosclerosis
* No thrombotic events within the past 6 months

Pulmonary:

* No aspirin-induced asthma

Other:

* No inability to take aspirin or clopidogrel bisulfate due to contraindications, allergies, or pre-existing medical conditions (e.g., active peptic ulcer disease or history of undiagnosed non-occult, non-hemorrhoidal gastrointestinal or other bleeding sources within the past 6 months)
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer that is currently in complete remission
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy and recovered
* No prior flavopiridol
* No more than 3 prior systemic chemotherapy regimens for recurrent or metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except oral contraceptives

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior surgery and recovered
* No prior carotid endarterectomy or other revascularization surgery

Other:

* No other concurrent antineoplastic therapies
* No active anticoagulation with INR 1.5 or greater
* No low-molecular weight heparin or equivalent
* Concurrent bisphosphonates for calcium maintenance allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Conley, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Center for Cancer Research, Bethesda, Maryland